CLINICAL TRIAL: NCT01746966
Title: US Investigation of Gleno-humeral Joint by Anterior Access With Measurement of Rotator Interval in Patients With Rheumatoid Arthritis and Healthy Controls
Brief Title: Anterior Shoulder US - a New Access
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: 0260-10CTIL
Record Dates: First submitted 2012-11-22; First posted 2012-12-11 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Rheumatoid Arthritis
Keywords: gleno-humeral joint synovitis; anterior shoulder US; rotator interval
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Rheumatoid Arthritis: 20 patients age of 20-60 with Rheumatoid Arthritis according to ARA 1987 revised criteria and disease activity Disease Activity Score (DAS) 3-5
- Healthy controls participants: Healthy controls age of 20-60 according to conclusion of preventive medicine department

SUMMARY:
1. Investigate Gleno-Humeral Joint (GHJ) by anterior approach:

   A - Measurement of GHJ thickness at 3 points and average value calculation on body supine position and with arm supinated, maximal externally rotated with elbow angle 90 degrees
   * By longitudinal access with transducer position laterally to coracoids along to the GHJ line, located as diagonal form lower to forward and lateral direction with demonstration the joint cartilage posteriorly and subscapular tendon anteriorly (Fig.4)
   * By transversal access with 90 degrees to longitudinal and at 3 points: upper with coracoids visualization, middle and lower (Fig.5-7).

   B - Measurement of rotator interval with assessment of width and higher.
2. Comparison of the data with results of classic values have been received by posterior and inferior (axillar) approach.
3. Comparison of the results between patients with Rheumatoid Arthritis (RA) and healthy controls

DETAILED DESCRIPTION:
US scan was shown to be effective and useful for investigation of shoulder diseases. It is easy to implement and return, not expensive and not invasive, and precise for assessment. Glenohumeral joint is most inspected in elderly population. Most of shoulder syndromes are not related to joint diseases, but to adjacent tissue problem. However, US is preferred method for assessment GHJ by rheumatologists. But inflammatory changes in GHJ found limited attention in medical imaging literature. So far there is assessment of GHJ synovitis with disclosure of synovial fluid and pannus in subdeltoid (subacromial) bursa and biceps tendon, connected to GHJ space, by axillar and posterior access. Subdeltoid bursitis and biceps tenosynovitis are common used for inflammatory assessment of the shoulder. Anterior approach for GHJ assessment has not been used before our last trial. A problem of patients with synovitis in GHJ is difficulties to pick up shoulder to lateral side (abduction) till 90 degrees for axillar approach. We proposed anterior access for GHJ synovitis assessment. Certain position of the shoulder and measured data of healthy controls enabled diagnostic of GHJ synovitis with minimal movement of ill shoulder. In other report we showed US differences between GHJ and subscapular tendon on the anterior approach. These two publications showed anterior shoulder US in sitting position with arm externally rotated and supinated. We should recognize problems of these trials related to wrong identification of GHJ space. As we realized later this incorrect detection was associated with missing two orienteer structures: GHJ cartilage located behind and subcscapular tendon situated forward to GHJ space. From our present view, these two criteria are corn stone for GHJ visualization. Because lack obvious picture of these 2 structures GHJ demonstration is unclear and exposed to confusion with subscapular tendon. Moreover, our further experience of multiple anterior US studies showed that presentation of GHJ in position for supination and external rotation in sitting position is associated with poor visualization of GHJ cavity. The reason is position of GHJ to be hidden behind humeral head due to differences between round humeral head and oval glenoid and twist GHJ structure forward-upper-laterally. Daily practice helped to resolve the problem. We found: a patient should be laid down supine, his elbow is bent to 90 degrees and the shoulder is rotated maximally externally. This condition is associated to fix shoulder girdle, glenoid move anteriorly, humeral head move posteriorly, and much more complete external shoulder rotation is achieved opening GHJ for investigation. Shoulder CT shows that glenoid surface is in plane open to upper, forward and lateral side. It obligates to turn of transducer according to direction of investigated joint placed along the glenoid surface. That means, longitudinal study of GHJ requests transducer position under certain angle along to joint line. Transversal study is implemented under angle 90 degree to the joint line. Other problem is that synovitis may developed at early stage only within limited region of the joint and in region much more susceptible to inflammation and dilatation, like that rotator interval: anterior upper region which is covered only by the joint capsule with lower resistance to distention. That region is referred as rotator interval, a distance between supraspinatus (laterally) and subcapularis (medially) tendons attachment, when shoulder supinated and externally rotated. This region has been recently used for synovial biopsy.

Materials and methods:

US will be performed for 20 healthy controls and 20 patients with RA. US scan will be fulfilled symmetric both sides. Diagnosis RA is relied on anamnesis data, physical examination, and laboratory findings. Synovial swelling, synovial tenderness, local fever of joint region, active and passive limitation, accelerated erythrocyte sedimentation rate(ESR) upper 40mm/hr (N<12), C reactive protein (CRP) upper 1.5mg/dl (N<0.5) were clinical signs of active inflammation. Twenty healthy controls did not complain of shoulder pain and limitation and their physical examination was unremarkable.

Study process:

US scan will be performed as prospective study for 20 healthy controls from department of preventive medicine and for 20 patients with RA age of 20-60 by to classic approaches: posterior and inferior and new anterior access. The last was accompanied by measurement of GHJ space and rotator interval in upper limb position of supination and external rotation. Comparison will be implemented between data of different positions and RA patients compared with controls.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy controls age of 20-60 according to conclusion of preventive medicine department
2. Patients with RA according to ARA 1987 revised criteria and disease activity DAS 3-5

Exclusion Criteria:

1. Past shoulder trauma
2. Shoulder osteoarthritis
3. Rotator cuff disorders
4. Shoulder injections
5. Cervical spondylosis with nerve root compression, Cervical symptomatic disc syndromes

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 20 healthy controls from department of preventive medicine and 20 patients with Rheumatoid Arthritis age of 20-60
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2012-12; Primary Completion 2015-06 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Measurement of GHJ thickness and of rotator interval | Six months
  A - Measurement of GHJ thickness at 3 points and average value calculation on body supine position and with arm supinated, maximal externally rotated with elbow angle 90 degrees
  * By longitudinal access with transducer position laterally to coracoids along to the GHJ line, located as diagonal form lower to forward and lateral direction with demonstration the joint cartilage posteriorly and subscapular tendon anteriorly (Fig.4)
  * By transversal access with 90 degrees to longitudinal and at 3 points: upper with coracoids visualization, middle and lower (Fig.5-7).
  B - Measurement of rotator interval with with assessment of width and higher.

SECONDARY OUTCOMES:
Data of comparison between measurement of GHJ in anterior and axillar access and anterior and posterior access in patients with Rheumatoid Arthritis and Controls. | Eight months
Data of comparison in measurement of rotator interval in patients with Rheumatoid Arthritis and controls. | Eight months

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Rozin, MD, Principal Investigator — Rambam Health Care Campus and Technion
Locations (1):
- Rheumatology unit, Haifa, Israel